CLINICAL TRIAL: NCT05974800
Title: Identification of Potential Improvements in the Acute Care Pathway for Cancer Patients in the Emergency Department (OVERSEE - II Trial)
Brief Title: Potential Improvements in Emergency Department Care for Cancer Patients According to Clinical Staff
Acronym: OVERSEE-II
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Jason den Duijn, Principal Investigator, Erasmus Medical Center
Other Study IDs: 10842
Record Dates: First submitted 2023-07-18; First posted 2023-08-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-08

CONDITIONS: Cancer; Emergencies
MeSH Terms: conditions — Neoplasms; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cancer patients: All adult patients with solid or hematological malignancies and receiving systemic therapy or having received systemic therapy within the last 3 months that are admitted to the emergency department of the Erasmus medical center for the oncology, hematological, lung- and neuro-oncology medical unit are eligible for inclusion.
  Interventions: Behavioral: Emergency department caregivers interview

INTERVENTIONS:
Behavioral: Emergency department caregivers interview — The interview focuses on several parts of the emergency care process: The first part is regarding the actions that are executed during an emergency department visit. We will establish which actions are executed and why. The second part is regarding the suspected outcome for the patient. The third part will be about any potential improvements to the emergency care process for the patient.

SUMMARY:
The goal of this Single center prospective cross-sectional study is to identify the facilitators and barriers among caregivers in the emergency department that influence disposition of patients with solid and hematology malignancies. The main question it aims to answer is to categorize the facilitators and barriers identified by three groups of emergency department (ED) staff. Participants will be asked for permission, afterwards a short interview will be held with the different ED caregivers (ED nurse, attending physician and supervising physician).

DETAILED DESCRIPTION:
The goal of this to identify the facilitators and barriers among caregivers in the emergency department (ED) that influence disposition of patients with solid and hematology malignancies. Participants will be asked for permission, afterwards a short interview will be held with the different caregivers (ED nurse, attending physician and supervising physician) in the ED. The interviews will be held in the order of the ED care pathway, meaning ED nurse first, treating physician second and supervising physician at last. The interviews will be conducted for every patient with each of the caregivers. Each interview will be conducted after the caregiver has made the first examination of the patient. The interview focuses on several parts of the emergency care process: The first part is regarding the actions that are executed during an ED visit. We will establish which actions are executed and why. The second part is regarding the suspected outcome for the patient. The third part will be about any potential improvements to the emergency care process for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid or hematological malignancies and receiving system therapy or having received systemic therapy within the last 3 months.
* Presented at or admitted from the emergency department for the oncology, hematology, neuro- or lung-oncology clinical unit.
* Awake and conscious.
* Possible to answer questions within the same shift / day after presentation in the ED.

Exclusion Criteria:

* <18 years old.
* Only received a surgical intervention as cancer treatment.
* Not willing or able to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the emergency department (ED) of Erasmus medical center (MC) yearly around 1600 patients with cancer are presented to the ED. Based on the study design we will conduct interviews with 75 to 100 patients with solid and hematologic malignancies, who are receiving systemic therapy or have received systemic therapy within the last 3 months and are admitted to the ED department of the Erasmus MC for the oncology, hematology, lung- and neuro-oncology medical unit. If present, the interview will also be held with the family caregiver.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Clusters of facilitator and barriers identified by the emergency department (ED) nurse | Through study completion, an average of 6 months
  (Sub)Clusters of facilitator and barriers identified by the ED nurse for the ED care of patients with cancer
Clusters of facilitator and barriers identified by the treating physician | Through study completion, an average of 6 months
  (Sub)Clusters of facilitator and barriers identified by the treating physician for the ED care of patients with cancer
Clusters of facilitator and barriers identified by the supervising physician | Through study completion, an average of 6 months
  (Sub)Clusters of facilitator and barriers identified by the supervising physician for the ED care of patients with cancer

SECONDARY OUTCOMES:
Emergency department (ED) length of stay (LOS) | Through study completion, an average of 6 months
  Emergency department length of stay
Disposition | Through study completion, an average of 6 months
  Outcome after ED admission, being home or admission
Correlation between ED-LOS and disposition | Through study completion, an average of 6 months
  Correlation between ED-LOS and disposition
Years of medical experience | Through study completion, an average of 6 months
  Number of years a medical staffmember is working in health care
Need for imaging | Through study completion, an average of 6 months
  Was imaging ordered during ED visit and which kind
ED nurse agreement of disposition | Through study completion, an average of 6 months
  Agreement between ED nurse expected disposition and the actual disposition
Attending physician agreement of disposition | Through study completion, an average of 6 months
  Agreement between treating physician expected disposition and the actual disposition
Supervising physician agreement of disposition | Through study completion, an average of 6 months
  Agreement between supervising physician expected disposition and the actual disposition
Time-to-disposition | Through study completion, an average of 6 months
  The time between patient's arrival at the ED and the decision to disposition
Time-to-ward | Through study completion, an average of 6 months
  The time between the decision to hospitalize and the arrival at the ward
Correlation between time-to-disposition and the ED-LOS | Through study completion, an average of 6 months
  Correlation between time-to-disposition and the ED-LOS
Correlation between time-to-ward and the ED-LOS | Through study completion, an average of 6 months
  Correlation between time-to-ward and the ED-LOS
Difference in categories | Through study completion, an average of 6 months
  The difference in the percentages in categories between the different caregivers
ED nurse summary of actions | Through study completion, an average of 6 months
  Summary of actions taken by ED nurse in the ED care for patients with cancer
Attending physician summary of actions | Through study completion, an average of 6 months
  Summary of actions taken by attending physician in the ED care for patients with cancer
Supervising physician summary of actions | Through study completion, an average of 6 months
  Summary of actions taken by supervising physician in the ED care for patients with cancer
ED crowding | Through study completion, an average of 6 months
  Degree of crowding in the ED, consisting of number of patients in the ED and the ED crowding color code
Difference in clusters per group between day, evening and night | Through study completion, an average of 6 months
  Difference in clusters per ED staff group between day, evening and night
Difference in clusters per group between weekdays and weekend | Through study completion, an average of 6 months
  Difference in clusters per group between weekdays (Monday 08:00 till Friday 16:00) and weekend (Friday 16:01 till Monday 7:59)

OTHER OUTCOMES:
Patient characteristics | Through study completion, an average of 6 months
  age, sex, type of cancer, type of treatment, main complaint, triage category, number of prior ED visits.

CONTACTS AND LOCATIONS:
Overall Officials: Jason den Duijn, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No